CLINICAL TRIAL: NCT01069055
Title: Pre-emptive Intravenous Analgesia for Elective Inguinal Hernia Repair: Prospective Randomized Double-blinded Placebo Controlled Comparison of Lornoxicam and Paracetamol
Brief Title: Comparison of Lornoxicam and Paracetamol for Pre-emptive Intravenous Analgesia for Elective Inguinal Hernia Repair
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Diskapi Teaching and Research Hospital, Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HerniaAnalgesia2010-001
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Inguinal Hernia; Postoperative Pain
Keywords: inguinal hernia; surgery; general anesthesia; analgesia; pre-emptive; SF36
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Control (Placebo Comparator): Group I (Placebo Control) 100 ml intravenous saline infusion as placebo 30 minitues before the surgery.
  Interventions: Other: Sterile Saline
- Lornoxicam (Active Comparator): Group II: 8 mg intravenous lornoxicam infusion in 100 ml saline 30 minitues before the surgery.
  Interventions: Drug: Intravenous lornoxicam
- Paracetamol (Active Comparator): Group III: 1 g intravenous paracetamol infusion in 100 ml saline 30 minitues before the surgery.
  Interventions: Drug: Intravenous paracetamol

INTERVENTIONS:
Other: Sterile Saline — Group I: 100 ml intravenous saline infusion as placebo 30 minitues before the surgery.
  Other Names: Saline
  Arms: Placebo Control
Drug: Intravenous lornoxicam — Group II: 8 mg intravenous lornoxicam infusion in 100 ml saline 30 minitues before the surgery.
  Other Names: Lornoxicam: Xefo
  Arms: Lornoxicam
Drug: Intravenous paracetamol — Group III: 1 g intravenous paracetamol infusion in 100 ml saline 30 minitues before the surgery.
  Other Names: Paracetamol: Perfalgan
  Arms: Paracetamol

SUMMARY:
The purpose of this study is to determine whether lornoxicam or paracetamol is more effective in providing pre-emptive analgesia for adult patients undergoing elective unilateral inguinal hernia repair under general anesthesia.

DETAILED DESCRIPTION:
Early postoperative pain is the major cause that may restric physical activity of the patients and delay in returning work. Newer non-steroid analgesic drugs (NSAD) can be helpful in overcoming this problem, especially in pre-emptive use. In this prospective randomized placebo controlled double blinded study we aimed to determine whether lornoxicam, as a NSAD, or paracetamol is more effective in providing pre-emptive analgesia for patients undergo elective unilateral inguinal hernai repair under general anesthesia. 60 patients above the age of 18, ASA score of I to III will be assigned into 3 groups. All the patients will be operated under general anesthesia. Recurrent hernia cases, pregnant or lactated women, patients allergic to the two drugs, patients with documented gastric disorders or bleeding disorder or under anticoagulent therapy will be excluded.

Group designs:

Group I: 100 ml intravenous saline infusion as placebo 30 minitues before the surgery.

Group II: 8 mg intravenous lornoxicam infusion in 100 ml saline 30 minitues before the surgery.

Group III: 1 g intravenous paracetamol infusion in 100 ml saline 30 minitues before the surgery.

All patients will receive patient controlled intravenous analgesia with morphine for 24 hours postoperatively.

Postoperative pain levels will be determined by VAS (visual analog scale) and morphine consumption will be recorded.

Patients will be prescribed with oral paracetamol (300 mg) plus codein (15 mg)at discharge at the end first 24 hours.

Patients will be asked to record daily consumption of given analgesic, pain response to physical activity by using Likert scale, and VAS scores daily.

The first follow-up examination will take place on day-7. The patients will be asked to keep recording the same parameters until the second hospital visit at 4th week.

On the follow-up examination at 4th week quality of life will be determined by SF-36 form.

The results will be analyzed using SPSS for Windows software.

ELIGIBILITY:
Inclusion Criteria:

* inguinal hernia
* unilateral hernia
* general anesthesia
* elective repair

Exclusion Criteria:

* drug allergy
* bilateral hernia
* local anesthesia
* local blockade
* regional anesthesia
* emergency surgery
* complicated hernia
* recurrent hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain and comfort | 24 and 48 hours

SECONDARY OUTCOMES:
Postoperative late pain complaint and quality of life | 4. week

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Sonmez, MD, Principal Investigator — Diskapi Teaching and Research Hospital
Locations (1):
- Diskapi Teaching and Research Hospital, Ankara, Turkey (Türkiye)